CLINICAL TRIAL: NCT05778162
Title: Evaluation of the Usability and Clinical Utility of the Synovasure® RISC Panel
Brief Title: RISC Panel Remnant Sample Collection
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: DTU2022-21DI
Record Dates: First submitted 2023-01-23; First posted 2023-03-21 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2024-12

CONDITIONS: Arthritis, Inflammatory
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The study will collect synovial fluid remnant samples from up to 1000 patients with a painful and/or swollen knee(s) for which arthrocentesis is performed as part of the patient's standard of care. De-identified leftover remnant samples will be frozen for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Synovasure® RISC™ Panel — The Synovasure® RISC™ Panel is a laboratory-developed test (LDT) panel (CD Laboratories, Clinical Laboratory Improvement Amendments [CLIA] Registration No.: 21D0216863) intended to provide indications for diagnosing different types of arthritis that may correspond to higher risk levels for postoperative complications in patients experiencing knee pain and/or inflammation prior to primary knee arthroplasty.

SUMMARY:
The primary objective of this study is to evaluate the usability and clinical utility of the Synovasure® RISC™ Panel.

The secondary objective of this study is to create a repository of well-characterized synovial fluid samples from patients with knee pain and/or inflammation to be used for future research.

DETAILED DESCRIPTION:
The Synovasure® RISC Panel™ constitutes a single source of pre-operative biomarker testing with high predictive value for the diagnosis of single or multiple arthritis conditions, that may correspond to a relative level of inflammation and post-operative complication and infection risk in patients with knee pain and/or inflammation.

The aim of this clinical performance post-market clinical follow-up (PMCF) study is to evaluate the usability and clinical utility of the Synovasure® RISC Panel™ using comparative analyses between the suspected diagnosis, patient demographics, conditions, symptoms, medical history and the Synovasure® RISC Panel™ results. The secondary objective of this study is to create a repository of well-characterized synovial fluid samples from patients with knee pain and/or inflammation to be used for future research.

Investigators will perform arthrocentesis as part of the patient's standard of care. Remnant samples will be transferred in the tubes included with the Synovasure® Arthritis Specimen Transportation kit, in accordance with instructions and the requisition form. Additional case report forms (CRFs) to collect demographic, and clinical data beyond what is included in the requisition form and the Panel results accession identification (ID) will be provided. Sample collection and shipment to CD Laboratories (CDL) may be limited to Monday-Wednesday. A maximum of three samples per transportation kit will be shipped as soon as the samples are collected. CDL will perform RISC™ Panel testing and identifiable results will be provided to enable the centers to pair the test results with clinical outcome data. De-identified leftover remnant samples will be frozen and all data, including any available clinical outcome data, will also be entered into a de-identified database of results and made accessible to all participating investigators for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee pain and/or inflammation and planned arthrocentesis

Exclusion Criteria:

* Patient is unwilling or unable to give oral consent
* Patient has any condition that would, in the judgment of the Investigator, place the patient at undue risk or interfere with the study
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant)
* Patient had an arthrocentesis of the index joint less than 2 weeks from the planned arthrocentesis
* Insufficient synovial fluid sample of < 1.5 mL
* Patient age < 18 or > 89

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients experiencing knee pain and/or inflammation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Rate of agreement | 2 years
  This study is intended to characterize the performance of the Synovasure® RISC™ Panel in a real-world environment. The primary endpoint of this study is the rate of agreement (positive and negative) of the test result with the suspected diagnosis. The suspected diagnosis of the index knee will be collected prior to the Synovasure® RISC™ Panel analyses to be subsequently matched to the Synovasure® RISC™ Panel results.

SECONDARY OUTCOMES:
Relationship between patient characteristics and panel results | 2 years
  The secondary endpoint will consist of an exploration of potential correlations between the subject characteristics and results of the RISC panel diagnostics. Analysis of Variance (ANOVA) will be used to test for associations, while chi-square tests or Fisher's exact tests will be used for categorical variables. Logistic regressions may be performed to examine diagnostic accuracy based on variables identified to be significant predictors (p-value ≤ 0.05) from the univariate analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Toler, Study Director — Zimmer Biomet
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided